CLINICAL TRIAL: NCT02168569
Title: In Vivo Efficacy of Artemether-lumefantrine and Amodiaquine-artesunate for the Treatment of Uncomplicated Falciparum Malaria in Children: A Multisite, Open-label, Two-cohort Clinical Trial in Mozambique.
Brief Title: In Vivo Efficacy of Artemether-lumefantrine and Amodiaquine-artesunate in Mozambican Children
Acronym: MEFI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Investigacao em Saude de Manhica (Other)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 134/CNBS/11
Record Dates: First submitted 2014-06-13; First posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Malaria
Keywords: treatment; artemisin-based combinations; children
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; amodiaquine, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Active Comparator): 5 sites, namely Manhiça, Dondo, Montepuez, Tete and Chokwe
  Interventions: Drug: Coartem™ (Artemether-lumefantrine combination)
- Cohort 2 (Active Comparator): 3 sites, namely Montepuez, Dondo and Chokwe
  Interventions: Drug: Coarsucam™ (Amodiaquine-artesunate combination)

INTERVENTIONS:
Drug: Coartem™ (Artemether-lumefantrine combination) — AL (Coartem™) was administered twice daily for three days (six doses in total) with dosage determined according to body weight: one tablet (20mg artemether and 120mg lumefantrine) for children 5 to <15kg, two tablets per dose for those 15 to <25kg, and three tablets per dose for those 25 to <35kg.
  Arms: Cohort 1
Drug: Coarsucam™ (Amodiaquine-artesunate combination) — AQ-AS (Coarsucam™) was administered once daily according to body weight: one 25mg artesunate and 67.5mg amodiaquine tablet in children <9kg, one 50mg artesunate and 135mg amodiaquine tablet in children 9-17.9kg; and one 100mg artesunate and 270mg amodiaquine tablet in children >18-35kg.
  Arms: Cohort 2

SUMMARY:
This is a classical in vivo clinical trial, following World Health organization's recommendations, ran as a multisite study within Mozambique trying to assess the efficacy and safety in 5 sites of the two oral ACTS artemether-lumefantrine (AL) and Amodiaquine-Artesunate (AQ-AS), first and second line treatment for malaria in mozambique, respectively, for the treatment of uncomplicated malaria in children aged<5 years.

DETAILED DESCRIPTION:
This study followed WHO recommendations for in vivo antimalarial efficacy trials.

The study population comprised children aged 6 to 59 months with microscopically confirmed acute uncomplicated malaria. Other inclusion criteria included body weight ≥5kg, the presence of fever (≥37.5°C axillary) or a history of fever in the preceding 24 hours, P. falciparum malaria mono infection with an asexual blood density ≥2,000/µL and <200,000/µL, and the absence of severe signs of complicated malaria as defined by WHO. Key exclusion criteria included mixed malarial infections, haemoglobin <5g/dL, severe malnutrition, intake of anti-malarials within the preceding seven days, ongoing prophylaxis in HIV positive patients with cotrimoxazole or the intake of any other drug with anti-malarial activity, and any serious underlying disease. Patients satisfying the inclusion criteria were enrolled if the parent/guardian signed a detailed written informed consent.

Eligible patients were consecutively assigned to the cohort and treated with AL (cohort 1) or AQ-AS (cohort 2). AL (Coartem™) was administered twice daily for three days (six doses in total) with dosage determined according to body weight: one tablet (20mg artemether and 120mg lumefantrine) for children 5 to <15kg, two tablets per dose for those 15 to <25kg, and three tablets per dose for those 25 to <35kg. AQ-AS (Coarsucam™) was administered once daily according to body weight: one 25mg artesunate and 67.5mg amodiaquine tablet in children <9kg, one 50mg artesunate and 135mg amodiaquine tablet in children 9-17.9kg; and one 100mg artesunate and 270mg amodiaquine tablet in children >18-35kg. All treatments were directly observed for a minimum of 30 minutes. Vomiting occurring within the first 30 minutes implied the repetition of the full dose of treatment. For those patients living far away from the health facilities, and for which direct observation of the evening doses of AL was challenging, admission was offered for the first three days of the study.

Antipyretics, such as paracetamol, were used to control fever>=38ºC. In the event of severe malaria or danger signs, the patient was hospitalized and received intravenous quinine, according to the national malaria treatment policy. Rescue therapy according to national malaria treatment guidelines was also administered in cases of early or late treatment failure

Follow-up visits took place on days 1, 2, 3, 7, 14, and 28 after enrolment or at any time point whenever the child was sick. Patients who prematurely discontinued either study drug or the study were excluded from the study. Vital signs and body temperature were assessed during each follow-up visit. Adverse events were recorded and assessed for severity and association with study medication.

Thick and thin Giemsa-stained blood slides were prepared before each dose was administered and at every follow-up visit of days 2, 3, 7, 14, 21 and 28. Slides were examined by two independent microscopists and considered negative if no parasites were seen after examination of 200 oil-immersion fields in a thick blood film. Species determination (and thus conformation of monoinfection) was made based on assessment of thin films. Blood samples for PCR analysis were collected from every patient at baseline and at days 7, 14 and 28, day of treatment failure or at any other unscheduled visit. PCR was performed centrally for all cases of recurrent parasitaemia from day 7 onwards to distinguish recrudescence from reinfection according to the standardized WHO method

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 to 59 months
* Weight Greater than or equal to 5 kg
* Absence of severe malnutrition;
* Mono-infection with Plasmodium falciparum in blood, confirmed by microscopy;
* Parasite density between 2,000 and 200,000 asexual parasites per microliter of blood;
* Axillary temperature ≥ 37.5 C° or history of fever in the last 24 hours;
* Lack of danger signs, or no signs of severe and / or complicated malaria according to the WHO definition
* Ability to swallow the drugs
* Haemoglobin greater than 5.0 g / dl
* Residents within the study area and have the possibility of an adequate follow-up in the days of monitoring for a period of 28 days;
* Absence of a history of hypersensitivity to study medications;
* Informed consent of parents, guardians or caregivers (legal guardian) after explaining the purpose of the study.

Exclusion Criteria:

* Presence of any danger sign or severe or complicated Plasmodium falciparum malaria according to WHO definitions
* Presence of fever due to diseases other than malaria (eg measles, acute respiratory infection, severe diarrhea with dehydration) or other known diseases, with chronic or serious illnesses (cardiac, renal, hepatic or known infection with HIV AIDS),
* Presence of severe malnutrition (defined as a child whose growth pattern is below the 3rd percentile, mid-upper-arm circumference <110mm, weight / height <70% according to the WHO tables, or the presence of bilateral edema of the lower limbs)
* Multi or mono-infection by another Plasmodium species detected by microscopy;
* Regular medication that may interfere with the pharmacokinetics of antimalarials;
* History of hypersensitivity or contraindication to study drug;
* A history of taking antimalarial drugs or drugs with antimalarial activity in less than 7 days.
* Continuous prophylaxis with cotrimoxazole in HIV positive children

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To measure the Day 28, PCR corrected cure rates of artemether-lumefantrine (Coartem) and Amodiaquine-artesunate (Coarsucam). | 28 days
  This cure rate is defined as the proportion of patients with adequate clinical and parasitological response (ACPR) at Day 28, once PCR correction to differentiate recrudescences friom new infections have been applied (and hence only considering as treatment failures those parasite recurrences confirmed as recrudescences).

SECONDARY OUTCOMES:
to evaluate the incidence of adverse events | 28 days
  To evaluate the incidence of adverse events, including the variation of haemoglobin levels throughout follow-up, during the 28 days that each subject will be followed
PCR uncorrected Day 28 efficacy of AL and AQ-AS | 28 days

CONTACTS AND LOCATIONS:
Locations (5):
- Mozambique (5):
  - Hospital Rural de Montepuez, Montepuez, Cabo Delgado Province
  - Hospital Rural de Chókwe,, Chokwé, Gaza Province
  - Centro de Investigação em Saúde de Manhiça, Manhiça, Maputo Province
  - Centro de Saúde de Dondo, Dondo, Sofala
  - Hospital Provinvial de Tete, Tete, Tete